CLINICAL TRIAL: NCT07007026
Title: The Effectiveness of an Immersive Virtual Reality Intervention on Physical Fitness, Balance, Fall Risk, Fear of Falling, Fatigue, and Quality of Life in Geriatric Individuals
Brief Title: Effects of Immersive Virtual Reality on Physical Function, Fall-Related Outcomes, Fatigue, and Quality of Life in Older Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBF00-2024-0128
Record Dates: First submitted 2025-05-14; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Geriatric; Virtual Reality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Intervention (Experimental): In the virtual reality intervention group, older adults utilized an Oculus Meta Quest 2 headset (Meta Platforms, Inc., Menlo Park, CA, USA). The Meta Horizon application on the phone facilitated screen mirroring, enabling the observation of the task's progression by reflecting the headset screen. The FIT-XR application, available in the Oculus store, was utilized, and it offers a variety of exercise modes and interfaces, including options for in-door and outdoor scenarios. An exhaustive examination of all exercise modes within the application was conducted to enhance upper and lower extremity muscle strength, weight transfer, stepping, trunk control, endurance, coordination, cognitive functions, and the duration and difficulty level of the exercises. The evaluation process involved a meticu-lous assessment of the suitability of these exercises for elderly individuals. Consequently, the FIT-XR Boxing and FIT-XR Slam exercise modes were selected for utilization in the study.
  Interventions: Other: Immersive Virtual Reality
- Active Control Group (Active Comparator): A physiotherapist developed an exercise program for the control group, providing visual and detailed explanations appropriate for older adults and distributing brochures to participants. The participants were instructed to adhere to the exercise program thrice weekly for a period of eight weeks.
  Interventions: Other: Traditional Home-based Exercises

INTERVENTIONS:
Other: Immersive Virtual Reality — The intervention program was implemented over a period of eight weeks, with three ses-sions per week, each lasting 35 minutes.
  Arms: Virtual Reality Intervention
Other: Traditional Home-based Exercises — The participants were instructed to adhere to the exercise program thrice weekly for a period of eight weeks.
  Arms: Active Control Group

SUMMARY:
To investigate the effectiveness of an immersive virtual reality intervention on physical fitness, balance, physical activity level, risk of falling, fear of falling, fatigue, and quality of life in older adults compared to an active control group (ACG).

DETAILED DESCRIPTION:
This study aims to investigate the effects of virtual reality intervention on interrelated physical and psychosocial multidimensional parameters such as physical fitness, balance, fall risk, fear of falling, fatigue, and quality of life in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over 65 years of age
* Individuals with a Mini Mental Test score of 24 and above
* Individuals who can walk independently and do not use assistive devices
* Individuals who voluntarily agreed to participate in the study

Exclusion Criteria:

* Individuals diagnosed with neurological diseases (Stroke, Parkinson's, Multiple Sclerosis)
* Individuals with a diagnosis of cardiovascular disease (heart failure, endocarditis, myocarditis, cardiac arrhythmias) diagnosed with psychiatric or cognitive disorders
* undergone surgical operation in the last 6 months
* Visual impairment that makes it impossible for them to see virtual reality images
* Individuals diagnosed with vertigo, epilepsy
* Individuals diagnosed with cancer

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Balance | Assessments were conducted before the intervention and at the end of the 8-week inter-vention period. tment at 8 weeks
  Fullerton Advanced Balance Test is a test consisting of ten items in total, including standing with feet together and eyes closed, reaching forward by extending the arm to pick up an object (pen) held at shoulder level, turning 360 degrees in the right and left directions, stepping on and over 15 cm steps, tandem walking, standing on one leg, standing on foam with eyes closed, two-foot jump-ing, walking by turning the head, and reactive postural control. Each item is scored be-tween 0 and 4, with a maximum score of 40. A higher score indicates better balance ability and a lower score indicates poor balance ability.

SECONDARY OUTCOMES:
Physical Activity Level | Assessments were conducted before the intervention and at the end of the 8-week intervention period.
  The Physical Activity Scale for the Elderly (PASE) was used to assess the physical ac-tivity level of individuals. The scale evaluates the physical activity of elderly individuals in the last week. It includes leisure time activities, housework activities, and work-related physical activity components. It questions the amount of activities such as walking, light, moderate, vigorous sports and recreational activities, strengthening and endurance exercises, work-related activities such as walking and standing, light housework such as gardening and home repairs, and the amount of activities in the last week. The activities in the scale are evaluated according to the intensity and frequency of exercise: light, moderate, and heavy. Activity durations can be marked as less than 1 hour, between 1-2 hours, be-tween 2-4 hours and more than 4 hours. To calculate the total score, activity frequencies and activity weights are multiplied. The scores obtained for each activity are summed to ob
Physical Fitness | Assessments were conducted before the intervention and at the end of the 8-week intervention period.
  Senior Fitness Test includes a total of six functional tests assessing muscular strength, flexibility, aerobic endurance, balance and agility. 30-second sit and stand test was used to evaluate the muscle strength of the lower extremity and 30-second weight lifting test was used to evaluate the muscle strength of the upper extremity. Two-minute step test was used to assess aerobic endurance, which involves recording the total number of dominant side steps taken correctly for 2 minutes with a stopwatch. The chair sit-reach test was used to evaluate the flexibility of the lower extremity muscles and the back scratch test was used to evaluate the flexibility of the upper extremities. For the assessment of agility and dynamic balance, eight-step walk test was used, which involved getting up from the chair on com-mand, walking a distance of 2.44 meters without running but as fast as possible, and sit-ting back on the chair by turning around the cylinder ahead.
Risk of Falling | Assessments were conducted before the intervention and at the end of the 8-week inter-vention period. tment at 8 weeks
  Morse Falls Scale is a practical scale that can categorize patients according to their fall risk. It includes a total of six domains: pres-ence of a history of falls, presence of comorbidity, use of assistive devices, intravenous therapy status, transfer/walking and mental status. In the evaluation, fall risk is deter-mined with cut-off scores as suggested by Morse, with 0-24 points being the group with no fall risk, 25-50 points being the group with low fall risk, and 51 and above points being the group with high fall risk.
Fear of Falling | Assessments were conducted before the intervention and at the end of the 8-week intervention period.
  The International Fall Efficacy Scale (FES-I) is a scale consisting of a total of 16 items with each item ranging from 1-4 points. The mini-mum total score is 16 and the maximum score is 64. A high total score indicates a high fear of falling.
Fatigue | Assessments were conducted before the intervention and at the end of the 8-week intervention period.
  FACIT Fatigue Scale, which assesses the level of fatigue in the last seven days, was used to evaluate fatigue. It consists of 13 items in total, with each item scored between 0 and 4. The minimum total score is 0 and the maximum score is 52. The lower the total score, the higher the fatigue level of the individual.
Life Quality | Assessments were conducted before the intervention and at the end of the 8-week intervention period.
  World Health Organization Quality of Life Instrument-Older Adults Mod-ule(WHOQOL-Old) sensory functions, autonomy, past, present and future activities, so-cial participation, dying and death, and closeness are the 6 sub-domains and 24 items in total [46]. Each item is scored between 1 and 5 and a minimum of 4 and a maximum of 20 points can be obtained from each sub-domain. At the same time, the total score can be calculated by summing the score values. The maximum total score that can be obtained in the whole scale is 120 and the minimum total score is 24. The higher the total score, the higher the quality of life level of the individual.
Treatment Satisfaction | Assessments were conducted before the intervention and at the end of the 8-week intervention period.
  Visual Analog Scale consisting of a 100 mm long horizontal line was used for treat-ment satisfaction assessment. There are two descriptors at the beginning and end of the line indicating extreme satisfaction (not at all satisfied and very satisfied).
Virtual Reality Sickness | Assessments were conducted before the intervention and at the end of the 8-week intervention period.
  Virtual Reality Sickness Questionnaire (VRSQ) consists of two components, oculo-motor and disorientation, and 9 items in total.The items are scored on a 4-point scale ranging from 0 to 3 (0=none, 1=mild, 2=moderate, 3=very). The oculomotor impairment component consists of 4 items: general discomfort, fatigue, eye strain and difficulty focus-ing. The disorientation component consisted of 5 items: headache, head fullness, blurred vision, dizziness with eyes closed and vertigo. As a result of the questionnaire, oculomotor, disorientation and total scores are obtained. Oculomotor and disorientation scores are calculated by dividing the individual's component score by the total score obtained (as a percentage). The total score is calculated by the simple average method and a higher score indicates a higher level of movement disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Ender Angın Associate Professor Doctor, Study Director — Eastern Mediterranean University; Gözde İyigün Associate Professor Doctor, Study Director — Eastern Mediterranean University; Damla Parmak, Principal Investigator — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Mersin, Northern Cyprus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No